CLINICAL TRIAL: NCT06313658
Title: Enhancing Functional Hand Recovery Through Nerve Reconstruction in Total Brachial Plexus Birth Injury
Status: Recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Yousif Tarek El-Gammal, Assistant Lecturer, Assiut University
Other Study IDs: Total BPBI
Record Dates: First submitted 2024-03-02; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Brachial Plexus Injury
MeSH Terms: interventions — Plastic Surgery Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Total brachial plexus exploration and reconstruction — In the adopted strategy, anatomical reconstruction was always performed when feasible and the lower trunk was considered the primary reinnervation target. Anatomical reconstruction of the plexus was attempted in the presence of at least three available roots; the best quality root stump (usually C5) was used for hand reanimation, while the lower ruptured roots were directed towards the upper and middle trunks. If one or more of the remaining root stumps were of doubtful quality, the compromised roots were grafted to the posterior divisions of the upper and middle trunks, while elbow flexion could be restored by transferring the intercostal nerves (T3-5) to the lateral cord. The lateral root of the median nerve was also included in the intercostal nerve transfer to restore hand sensations. In all cases, the spinal accessory nerve was directly sutured to the suprascapular nerve to restore rotator cuff function.

SUMMARY:
Interpreting the published outcomes of hand function in total BPBI is confounded by a lack of clear documentation regarding detailed surgical findings and management strategies. Investigators have followed a well-defined protocol for surgical reconstruction with the primary objective being reinnervation of the lower trunk using the best available root. In this paper, Investigators outline the details of the strategy and provide a comprehensive analysis of the nerve reconstruction techniques and the resulting functional outcomes.

DETAILED DESCRIPTION:
Managing total BPBI cases is complex because surgical reconstruction must address the restoration of shoulder, elbow, and hand functions. In cases where multiple nerve root avulsions are present, prioritizing which functions to reinnervate shoulder, elbow, or hand becomes a critical decision. While attempts to restore hand function in adults with total brachial plexus lesions have yielded disappointing results, it has been shown that restoring hand function in infants with BPBI is more promising due to their enhanced neuro-regenerative capacities. Interpreting published outcomes of hand function in total BPBI is confounded by a lack of clear documentation regarding detailed surgical findings and management strategies. Various hand function scales that measure the individual joint movements or the global function of the hand and wrist have been used in the assessment of the outcomes, but none has quantitated the recovery of the intrinsic muscles of the digits or thumb. Furthermore, it is well-documented that the recovery of hand function can be a prolonged process, often extending up to eight years before reaching a plateau. The majority of the published studies have typically reported outcomes based on a minimum follow-up period of two years, which may not provide sufficient time to assess the full extent of hand function recovery.

Investigators have followed a well-defined protocol for the surgical reconstruction of total BPBI with the primary objective being restoration of hand function through reinnervation of the lower trunk followed by restoration of elbow and shoulder functions through innervation of the upper trunk. In this paper, Investigators outline the details of the surgical strategy and provide a comprehensive analysis of the nerve reconstruction techniques and the resulting functional outcomes. Furthermore, investigators explore and identify the factors that may significantly impact the recovery process.

ELIGIBILITY:
Inclusion Criteria:

* Patients Who underwent brachial plexus exploration and reconstruction for total OBPP.

who have reached at least four years of follow-up

Exclusion Criteria:

* Excluding children who had selective distal neurotization for restoration of specific functions without brachial plexus exploration or who had secondary procedures to the hand.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study will include at least 50 children:
  Who underwent brachial plexus exploration and reconstruction for total OBPP. who have reached at least four years of follow-up Excluding children who had selective distal neurotization for restoration of specific functions without brachial plexus exploration or who had secondary procedures to the hand.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-03-15 (Estimated); Primary Completion 2025-03-15 (Estimated); Study Completion 2025-03-15 (Estimated)

PRIMARY OUTCOMES:
Active Movement Scale (AMS) | 1 year
  All patients included in the study were evaluated using the Active Movement Scale (AMS), which grades upper extremity movements from 0 to 7. Scores of 6 or 7 would be considered successful in demonstrating functionally useful movement; this is a 50% and full range of movement against gravity, respectively.Attention was focused on sex movements primarily involving hand function including wrist, finger, and thumb flexion and extension.

SECONDARY OUTCOMES:
Al-Qattan pronation/Supination score | 1 year
  Separate assessments were performed of forearm pronation/supination as described by Al-Qattan
Raimondi hand score | 1 year
  Global hand function was assessed using the Raimondi scale; a score of 3 or more indicate a useful functional recovery

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospitals, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haerle M, Gilbert A. Management of complete obstetric brachial plexus lesions. J Pediatr Orthop. 2004 Mar-Apr;24(2):194-200. doi: 10.1097/00004694-200403000-00012. PMID 15076607
- [Background] Al-Qattan MM. Assessment of the motor power in older children with obstetric brachial plexus palsy. J Hand Surg Br. 2003 Feb;28(1):46-9. doi: 10.1054/jhsb.2002.0831. PMID 12531668
- [Background] Borschel GH, Clarke HM. Obstetrical brachial plexus palsy. Plast Reconstr Surg. 2009 Jul;124(1 Suppl):144e-155e. doi: 10.1097/PRS.0b013e3181a80798. PMID 19568147
- [Background] Pondaag W, Malessy MJ. Recovery of hand function following nerve grafting and transfer in obstetric brachial plexus lesions. J Neurosurg. 2006 Jul;105(1 Suppl):33-40. doi: 10.3171/ped.2006.105.1.33. PMID 16871868